CLINICAL TRIAL: NCT07222930
Title: Reactions to Learning Amyloid and Tau Results in Adults at Risk for Alzheimer's Dementia
Brief Title: Learning Amyloid and Tau Results
Status: Not yet recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0685; Protocol Version 12/10/25 (Other: UW Madison); SMPH/MEDICINE/GER-AD DEV (Other: UW Madison)
Record Dates: First submitted 2025-10-29; First posted 2025-10-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Amyloid; Tau; Alzheimer's Risk; dementia; biomarker testing; risk; pathophysiological changes; communication
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain; Dementia; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants from UW Alzheimer's Disease Research: Participants aged 50-89 who are cognitively unimpaired or have mild cognitive impairment will be enrolled from the Wisconsin Registry for Alzheimer's Prevention, Wisconsin Alzheimer's Disease Research Center Clinical Core, or other studies affiliated with the UW Alzheimer's Research Program.
  Interventions: Other: Disclose amyloid, tau results; Other: Follow-up Assessments

INTERVENTIONS:
Other: Disclose amyloid, tau results — Release of results from investigational agents conducted under IND 107114, IND 166860, and IND 134516
Other: Follow-up Assessments — self-report psychosocial and behavioral questionnaires

SUMMARY:
This is a prospective, single-cohort, single-center, observational study to assess if learning one's Alzheimer's disease biomarker test result impacts longitudinal psychosocial, behavioral, and neuropsychological outcomes, and to identify factors that moderate and mediate these outcomes. Participants enrolled in this study are requested to complete surveys at four timepoints after learning their Alzheimer's biomarker test results.

DETAILED DESCRIPTION:
The overall objective is to determine how learning one's amyloid and tau test results impacts longitudinal psychosocial, behavioral, and neuropsychological outcomes, and identify factors that moderate and mediate these outcomes.

The rationale is that by understanding factors that explain variability in reactions, biomarker communication and post-testing support can be tailored to optimize outcomes.

The central hypothesis is that learning biomarker profile will affect psychosocial, behavioral, and neuropsychological outcomes, and that these outcomes will be moderated by social determinants of health (SDOH) and perceived communication factors and mediated by illness perceptions and beliefs.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent.
* Willing to comply with all study procedures and be available for the duration of the study.
* Individuals at least 50 years of age.
* Enrolled in Wisconsin Registry for Alzheimer's Prevention (WRAP) or Alzheimer's Disease Research Center Clinical Core (ADRC)
* Previously adjudicated as cognitively unimpaired having mild cognitive impairment (MCI), or impaired but do not meet diagnostic criteria for mild cognitive impairment or dementia (classified as "Impaired-Not MCI" by the WRAP and ADRC cohorts) at their last WRAP or ADRC study visit at the time of enrollment into this study
* Have completed or able to complete amyloid and/or tau PET scans as part of a UW Alzheimer's Research Study

Exclusion Criteria:

* Diagnosis of dementia at the time of enrollment as determined by the most recent parent WRAP/ADRC study visit diagnostic consensus conference using standard NIA-AA 2011 diagnostic criteria. Participants who develop dementia after enrolling into this study may remain enrolled if they maintain decisional capacity and are able to follow study instructions and procedures.
* Individuals who lack decisional capacity to provide informed consent as determined by significant difficulty in understanding materials and information about study procedures during recruitment and/or informed consent discussions.
* Not suitable for study participation due to other reasons at the discretion of the investigators.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 240 participants aged 50-89 who are cognitively unimpaired or have mild cognitive impairment will be enrolled from the Wisconsin Registry for Alzheimer's Prevention, Wisconsin Alzheimer's Disease Research Center Clinical Core, or other studies affiliated with the UW Alzheimer's Research Program.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Impact of Neuroimaging in Alzheimer's Disease (INI-AD) Score | 1 month, 6 months, 12 months, 18 months
  Test-related distress will be assessed using the INI-AD instrument. Score range from 0-80 where higher scores indicate increased negative impact of test.
Stigma Impact Scale (SIS) Score | 1 month, 6 months, 12 months, 18 months
  Items are rated on a 4-point Likert scale ranging from strongly agree (4) to strongly disagree (1), and a fifth option of "not applicable" with higher total scores (24-96) indicating higher perceived stigma.
Control, Autonomy, Self-Realization, and Pleasure (CASP-12) | baseline, 1 month, 6 months, 12 months, 18 months
  This is a quality of life measure scored from 0-36 where higher scores mean better quality of life.
Future Time Perspective Scale | baseline, 1 month, 6 months, 12 months, 18 months
  Scores are from 1-7 where higher scores indicate higher engagement.

SECONDARY OUTCOMES:
Willingness to Prevent AD | baseline, 1 month, 6 months, 12 months, 18 months
  Willingness to seek clinical evaluation about brain health and AD risk will be assessed by the Willingness to Prevent AD Scale, 12 items on a 5-point scale are scored from 12-60 where higher numbers indicate an increased willingness to prevent AD. A sum score (or projected/comparable sum score for participants who complete less than 12 items) for items answered will be calculated as the mean multiplied by the total number of available items, to be comparable between participants who answer a different number of items.
Willingness to Prevent AD: Over the counter, prescription, clinical trial items | baseline, 1 month, 6 months, 12 months, 18 months
  Willingness to seek clinical evaluation about brain health and AD risk will also be assessed using 3 additional items added to the instrument, scored on a 5-point scale from 3-15 where higher numbers indicate an increased willingness to prevent AD.
Exercise Vital Sign Tool: Minutes per Week of Moderate or Vigorous Exercise | baseline, 1 month, 6 months, 12 months, 18 months
  Engagement in health behaviors will in part be assessed using the exercise vital sign tool. This is self-reported as number of days per week and average minutes per day of moderate to vigorous exercise (like a brisk walk). The number of days per week is multiplied by average minutes per day to compute the outcome of minutes per week of moderate or vigorous physical activity. .
Cognitive & Leisure Activity Scale (CLAS) | baseline, 1 month, 6 months, 12 months, 18 months
  Engagement in health behaviors will in part be assessed by the CLAS scale, scored from 0-80 where higher scores means increased participation in cognitive and leisure activities.
6-item questionnaire for Mediterranean diet | baseline, 1 month, 6 months, 12 months, 18 months
  Engagement in health behaviors will in part be assessed with the 6-item questionnaire for Mediterranean diet. Scores range from 0-6 with higher scores more closely resembling a Mediterranean dietary pattern.
Brief Pittsburgh Sleep Quality Index (B-PSQI) | baseline, 1 month, 6 months, 12 months, 18 months
  Engagement in health behaviors or willingness to engage in brain health behaviors, clinical trials, or treatments will in part be assessed using the B-PSQI, scored from 0-15 where higher scores indicate poorer sleep quality.
Number of Participants who Complete Advanced Directives | baseline, 1 month, 6 months, 12 months, 18 months
Clinical Trial Enrollment | baseline, 1 month, 6 months, 12 months, 18 months
  Clinical trial enrollment will be assessed using an item from the Willingness to Prevent AD survey that inquires about willingness and actual enrollment in clinical trials. Answers include: "will not do", "have not considered", "considered, but have not decided", "ready, will do", and "already did".
Communication Assessment Tool (CAT) Score | 1 month
  Communication will be assessed at the 1-month follow-up timepoint using CAT, scored from 15 to 75 where higher scores indicate better reported communication.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Clark, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored and shared back with the larger source studies (Wisconsin Registry for Alzheimer's Prevention and Wisconsin Alzheimer's Disease Research Center) to allow for investigators to request the data for future analyses.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified data will be available upon publication of related work or end of the project period, whichever comes first. Data will be preserved for at least five years following the end of the grant period.
Access Criteria: De-identified data can be requested by internal and external researchers through data request procedures set by the source studies.
URL: https://wrap.wisc.edu/data-requests-2/